CLINICAL TRIAL: NCT03138161
Title: SAINT: A Phase 1/2 Study of Safe Amounts of IPLIMUMAB, NIVOLUMAB and TRABECTEDIN for Previously Treated Advanced Soft Tissue Sarcoma (STS)
Brief Title: SAINT:Trabectedin, Ipilimumab and Nivolumab for Previously Treated Advanced Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sarcoma Oncology Research Center, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOC-1702
Record Dates: First submitted 2017-04-14; First posted 2017-05-03 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Advanced Soft Tissue Sarcoma; Metastatic Soft Tissue Sarcoma
Keywords: cancer immunotherapy, combination chemo-/immunotherapy
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin; Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase 1 (Experimental): Phase 1: 3-6 will be treated with escalating doses of Trabectedin every 3 weeks up to 18 doses. Dose Level 1 is 1.0 mg/m2; Dose Level 2,1.2 mg/m2; Dose Level 3,1.5 mg/m2. Beginning 2 weeks after the first dose of Trabectedin, all patients will be treated with Ipilimumab at 1 mg/kg every 12 weeks up to 5 doses, and Nivolumab at 3 mg/kg every 2 weeks up to 26 doses.
  Phase 2: All patients will be treated with the maximum tolerated dose of Trabectedin every 3 weeks. Beginning 2 weeks after the first dose of Trabectedin, all patients will be treated with Ipilimumab at 1 mg/kg every 12 weeks up to 5 doses, and Nivolumab at 3 mg/kg every 2 weeks up to 26 doses.
  Interventions: Drug: Trabectedin; Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Trabectedin — Trabectedinis an alkylating drug indicated for the treatment of patients with unresectable or metastatic liposarcoma or leiomyosarcoma who received a prior anthracycline-containing regimen.
  Other Names: Yondelis
Drug: Ipilimumab — Ipilimumab is a human cytotoxic T-lymphocyte antigen 4 (CTLA-4)-blocking antibody indicated for (1) treatment of unresectable or metastatic melanoma, and (2) adjuvant treatment of patients with cutaneous melanoma with pathologic involvement of regional lymph nodes of more than 1 mm who have undergone complete resection, including total lymphadenectomy.
  Other Names: Yervoy
Drug: Nivolumab — A fully human immunoglobulin (Ig) G4 monoclonal antibody directed against the negative immunoregulatory human cell surface receptor programmed cell death-1 (PD-1, PCD-1) with immune checkpoint inhibitory and antineoplastic activities. Nivolumab binds to and blocks the activation of PD-1, an Ig superfamily transmembrane protein, by its ligands programmed cell death ligand (PD-L1), overexpressed on certain cancer cells, and programmed cell death ligand (PD-L2), which is primarily expressed on APCs (antigen presenting cells). This results in the activation of T-cells and cell-medicated immune responses against tumor cells or pathogens. Activated PD-1 negatively regulates T-cell activation and plays a key role in tumor evasion from host immunity.
  Other Names: Opdivo

SUMMARY:
This is an open label, dose-seeking phase 1/2 study using escalating doses of TRABECTEDIN given intravenously with defined doses of IPILIMUMAB and NIVOLUMAB based on preliminary results of the Checkmate 012 trial for NSCLC (Hellman et al., 2016). For the Phase 1 Part of Study, only previously treated patients will be enrolled. For the Phase 2 Part of Study, previously treated patients will be enrolled.

DETAILED DESCRIPTION:
I. Dose Escalation Phase 1 of Study: The study will employ the standard "Cohort of Three" design (Storer, 1989). Three patients are treated at each dose level with expansion to six patients per cohort if DLT is observed in one of the three initially-enrolled patients at each dose level. If no DLT occurs after 2 doses, escalation to the next dose level will be permitted. The maximum tolerated dose is defined as the highest safely tolerated dose, where not more than one patient experienced DLT, with the next higher dose level having at least two patients who experienced DLT. Patients in the dose escalation study may continue treatment at their designated dose levels until disease progression or unacceptable toxicity occurs or up to 9 six-week cycles (one year) of therapy (up 18 TRABECTEDIN doses). No intra-patient dose escalation will take place.

Dose of IPILIMUMAB: 1 mg/kg IV over 30 min. q 12 weeks, beginning 2 weeks after first dose of TRABECTEDIN, until disease progression or unacceptable toxicity, up to 5 doses

Dose of NIVOLUMAB: 3 mg/kg over 30 min. q 2 weeks, beginning 2 weeks after first dose of TRABECTEDIN, until disease progression or unacceptable toxicity, up to 26 doses

Dose of TRABECTEDIN: Escalating doses of TRABECTEDIN IV as continuous intravenous infusion (CIV) over 24 hrs) q 3 weeks:

Dose Level I: 1 mg/m2 (n = 3-6); Dose Level II: 1.2 mg/m2 (n=3-6); Dose Level III: 1.5 mg.m2 (n=3-6)

II. Expansion Phase 2 of Study: Following dose escalation, an additional 22-28 previously untreated patients will receive TRABECTEDIN at the MTD and defined doses of IPILIMUMAB and NIVOLUMAB to assess overall safety and potential efficacy in a greater number of patients. Patients in the expansion phase of the study may continue treatment until significant disease progression (see criteria for discontinuation of therapy) or unacceptable toxicity occurs up to 9 six-week cycles (one year) of therapy.

Surgical Resection: After one or more treatment cycles, the principal investigator may recommend surgical debulking, complete surgical removal or a biopsy. If residual disease is present either by histopathological examination or by CT scan/MRI, repeat treatment cycles may be given 4 weeks after surgery, if the surgical incision has healed, and if the patient has < grade I toxicity.

Resected or biopsied tumors will be analyzed for the effects of this triple therapy on response, and immune cell trafficking in the tumor microenvironment. Fresh and paraffin embedded tissue blocks will be analyzed by FACS for PD-L1 and other biomarkers, including Tregs, CD8+, CD4+ cells etc. Immunohistochemistry for cyclin G1, cyclin D1 and Ki67 will be conducted to determine the tumor's proliferative state. Histopathologic examination for tumor necrosis and mitotic index will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet all of the inclusion criteria in order to be eligible to participate in the study, as follows:

  * Male or Female ≥ 18 years of age
  * Pathologically confirmed diagnosis of locally advanced unresectable or metastatic soft tissue sarcoma
  * For the Phase 1 Part of Study, previously treated patients will be enrolled. For the Phase 2 Part of Study, previously treated patients will be enrolled.
  * Ability to understand the purposes and risks of the study and has signed and dated a written informed consent form approved by the investigator's IRB/Ethics Committee
  * Willingness to comply with all study procedures and availability for the duration of the study.
  * Measurable disease by RECIST v1.1
  * ECOG performance status ≤1
  * Life expectancy of at least 3 months
  * Acceptable liver function: Bilirubin ≤ 1.5 times upper limit of normal (ULN; except subjects with Gilbert Syndrome who must have a total bilirubin level ≤ 3.0 ULN);AST (SGOT), ALT (SGPT) and alkaline phosphatase ≤ 3 x ULN (≤ 5 x ULN if liver metastases)
  * Acceptable renal function: Creatinine ≤1.5 times ULN or ≥ 60 mL/min (using the Cockcroft Gault formula)
  * Acceptable hematologic status (without hematologic support): WBC ≥2000/µL; ANC ≥ 1500 cells/μL; Platelet count ≥ 100,000/μL; Hemoglobin ≥ 9.0 g/dL; Normal PT, PTT, INR
  * All women of childbearing potential must have a negative pregnancy test and all subjects must agree to use highly effective means of contraception (surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 5 months for women and 7 months for men after the last dose.

Exclusion Criteria:

* All individuals meeting any of the exclusion criteria at baseline will be excluded from study participation, as follows:

  * Subjects with untreated CNS metastases. Subjects are eligible if CNS metastases have been adequately treated and have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to treatment initiation. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of ≤10 mg daily prednisone (or equivalent) for at least 2 weeks prior to treatment initiation.
  * Subjects with carcinomatous meningitis
  * Anticancer treatment with radiation therapy, chemotherapy, targeted therapy or other antitumor treatment within 2 weeks prior to study entry
  * Subjects who participated in an investigational drug or device study within 14 days prior to study entry
  * Females who are pregnant or breast-feeding
  * Unwillingness or inability to comply with the study protocol for any reason
  * Non-oncology vaccine therapy used for prevention of infectious disease within 4 weeks of trial enrollment
  * • History of or known or suspected autoimmune disease (exception(s): patients with vitiligo, Type I diabetes, resolved childhood atopic dermatitis, hypothyroidism, or hyperthyroidism that is clinically euthyroid at Screening are allowed). Other exceptions may be allowed following discussion with the Sponsor Medical Monitor for patients who have not received treatment for their autoimmune disorder in the past 3 years.
  * Systemic immunosuppression, including HIV positive status with or without AIDS
  * Skin rash (psoriasis, eczema) affecting ≥ 25% body surface area
  * Inflammatory bowel disease (Crohn's or ulcerative colitis)
  * Ongoing or uncontrolled diarrhea within 4 weeks of trial enrollment
  * Recent history of acute diverticulitis, intraabdominal abscess or gastrointestinal obstruction within 6 months of trial enrollment, which are known risk factors for bowel perforation
  * Patients with congestive heart failure or recent cardiac event
  * Evidence of severe or uncontrolled systemic disease or any other concurrent condition, including psychiatric, which in the principal investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the trial
  * Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
  * Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
  * Inadequate hematologic, renal or hepatic function defined by any of the following screening laboratory values: WBC ≤2000/µL; Neutrophils ≤1500/µL; Platelets ≤ 100,000/µL; hemoglobin ≤9.0 g/dL; Serum creatinine ≥1.5 x ULN or creatinine clearance ≤ 60 mL/min (using the Cockcroft Gault formula); AST/ALT ≥3 x ULN (≥ 5 x ULN if liver metastases); Total Bilirubin ≥1.5 x ULN (except subjects with Gilbert Syndrome who must have a total bilirubin level ≥ 3.0 ULN)
  * Current, active or previous history of heavy alcohol abuse
  * Pituitary endocrinopathy
  * Adrenal insufficiency or excess

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-04-13 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | 6 months
  Dose escalation study, determination of maximum tolerated dose (MTD) in previoiusly treated patients with soft tissue sarcoma followed by expansion to previously untreated patients with advanced STS

SECONDARY OUTCOMES:
Objective response rate (ORR), disease control rate (DCR) | 24 months
  Effect of triple therapy with trabectedin, ipilimumab and nivolumab on ORR and DCR in advanced soft tissue sarcoma
Progression free survival (PFS), 6 month PFS rate | 24 months
  Effect of triple therapy with trabectedin, ipilimumab and nivolumab on progression free survival (PFS), 6 month PFS rate
Overall survival (OS), 6 month OS rate | 24 months
  Effect of triple therapy with trabectedin, ipilimumab and nivolumab on overall survival in advanced soft tissue sarcoma

OTHER OUTCOMES:
Tumor response and PD-1, PD-L1 expression in tumors | 30 months
  Correlation of response with PD-L1 expression and other biomarkers in patients' tumors
Dexamethasone and immune related events | 30 months
  • Correlation of the timing and effect of dexamethasone use (necessarily given with TRABECTEDIN) on absolute lymphocyte count and the immune response, including immune related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Erlinda M Gordon, MD, Principal Investigator — Sarcoma Oncology Research Center
Locations (1):
- Sarcoma Oncology Research Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gordon EM, Sankhala KK, Chawla N, Chawla SP. Trabectedin for Soft Tissue Sarcoma: Current Status and Future Perspectives. Adv Ther. 2016 Jul;33(7):1055-71. doi: 10.1007/s12325-016-0344-3. Epub 2016 May 27. PMID 27234989
- [Background] Demetri GD, von Mehren M, Jones RL, Hensley ML, Schuetze SM, Staddon A, Milhem M, Elias A, Ganjoo K, Tawbi H, Van Tine BA, Spira A, Dean A, Khokhar NZ, Park YC, Knoblauch RE, Parekh TV, Maki RG, Patel SR. Efficacy and Safety of Trabectedin or Dacarbazine for Metastatic Liposarcoma or Leiomyosarcoma After Failure of Conventional Chemotherapy: Results of a Phase III Randomized Multicenter Clinical Trial. J Clin Oncol. 2016 Mar 10;34(8):786-93. doi: 10.1200/JCO.2015.62.4734. Epub 2015 Sep 14. PMID 26371143
- [Background] Hellman MD, Gettinger SN, Goldman JW, et al. CheckMate 012: Safety and efficacy of first-line (1L) NIVOLUMAB (nivo;N) and IPILIMUMAB (ipi;I) in advanced (adv) NSCLC. J Clin Oncol 2016, 34: (suppl; abstr 3001).
- [Background] Gordon EM, Sankhala KK, Stumpf N, Tseng WW, Chawla SP. Cancer immunotherapy with sequential administration of trabectedin and nivolumab in advanced soft tissue sarcoma. Presented at the Society of Immunotherapy for Cancer/ ITOC, Prague, Czech Republic, March, 2017